CLINICAL TRIAL: NCT02104934
Title: A Randomised Controlled Trial Comparing Single Shot Adductor Canal Block With Local Infiltration Analgesia for Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGHLIAACB2013
Record Dates: First submitted 2014-03-18; First posted 2014-04-07 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2015-07

CONDITIONS: Analgesia in Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Infiltration Analgesia (No Intervention): The Local Infiltration Analgesia group will receive local infiltration of ropivacaine 150mg, ketorolac 30mg, morphine 10mg, adrenaline 200mcg and vancomycin 500mg in a total volume of 75mls by the surgeon.
- Adductor Canal Block (Active Comparator): The Adductor Canal Block group of patients will receive intravenous ketorolac 30mg intra-operatively and an adductor canal block at the end of surgery. The block will be performed under real time ultrasound guidance and 30mls of 0.5% ropivacaine (150mg) is injected with a Stimuplex A100, 21G needle.
  Interventions: Procedure: Adductor Canal Block

INTERVENTIONS:
Procedure: Adductor Canal Block
  Arms: Adductor Canal Block

SUMMARY:
Total knee arthroplasty or replacement (TKA), a commonly performed surgery for osteoarthritis of the knee, is a painful procedure and requires a multimodal analgesic approach. A method for analgesia is local infiltration analgesia (LIA), where a mixture of drugs is injected around the knee joint.

Adductor canal block (ACB) is an alternative regional anaesthesia technique which has been shown to result in minimal thigh weakness.

The investigators aim to study if the analgesia provided by ACB is superior to LIA while preserving quadriceps strength.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary TKA under single shot spinal anaesthesia, between ages 45-85 years old, American Society of Anesthesiologists (ASA) physical status 1 to 3 and BMI 18-35 kg/m2

Exclusion Criteria:

* Patients unable to give consent, inability to communicate/ cooperate, patients with regular consumption of strong opioids (morphine, oxycodone) or steroids, allergy to local anaesthetics or any drugs included in the study, patients with lower limb surgery in the preceding year, patients with pre-existing neurological deficits and patients who have contraindications for spinal anaesthesia.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours | 24 hours
  morphine consumption in the first 24 hours (including morphine administered in recovery and via PCA).

SECONDARY OUTCOMES:
Pain Scores | 1, 6, 12, 24 hours; up to 48 hours postoperative
  Pain scores are recorded at 1, 6, 12, 24 and 48 hours post-operatively, assessed using a visual analog scale (0-100mm) at rest and during 45 degree passive flexion of knee.
Morphine Consumption | At 48 hours
  The balance usage after primary outcome
Postoperative Nausea and Vomiting | Up to 48 hours
  Presence/absence of nausea and vomiting, and total number of episodes of vomiting
Sedation Scores | Up to 48 hours
Quadriceps Strength | at 24 and 48 hours

OTHER OUTCOMES:
Presence of Complications | up to 48 hours
  Hematoma, wound infection, neurological deficits, any incidence of fall
Length of Hospital Stay | Up to 30 days
  Number of days till discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yean Chin Lim, MBBS, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided